CLINICAL TRIAL: NCT05689476
Title: Evaluation of the Relationship Between Electrical Activity of the Diaphragm and Respiratory Mechanics During Neurally Adjusted Ventilatory Assist in Lung Transplant Patients and in Patients Affected by Acute Respiratory Failure.
Brief Title: Electrical Activity of the Diaphragm and Respiratory Mechanics During NAVA
Acronym: NAVAMECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAVAMECH
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-01

CONDITIONS: Work of Breathing; Lung Transplantation; Neurally Adjusted Ventilatory Assist; Ventilator-Induced Lung Injury; Acute Respiratory Failure (ARF)
Keywords: Lung Injury; Ventilator-Induced Lung Injury; Neurally Adjusted Ventilatory Assist
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Lung Injury

STUDY DESIGN:
Masking Description: none (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NAVA group (Experimental): Nava ventilation
  Interventions: Device: NAVA GROUP

INTERVENTIONS:
Device: NAVA GROUP — NAVA ventilation: Assisted Ventilation Mode, synchronized, through EAdi catheter, with patient's inspiratory effort and proportional to respiratory drive

SUMMARY:
Protective ventilatory strategy should be applied to reduce ventilator-induced lung injury (VILI) after Lung Transplantation (LTx) or in case of acute respiratory failure requiring invasive mechanical ventilation. Neurally Adjusted Ventilatory Assist (NAVA) is an assisted ventilation mode in which respiratory support is coordinated by the electrical activity of the diaphragm (EAdi). Aim of the study is to assess the physiological relationship between neural respiratory drive, as assessed by EAdi, and tidal volume, driving pressure, and mechanical power, at different levels of ventilatory assist, in the absence of pulmonary vagal afferent feedback or during acute respiratory failure. Additional parameters will be collected: Pmus, Pocc, transpulmonary pressure etc.

DETAILED DESCRIPTION:
Lung transplantation (LTx) is an important treatment option for select patients with end-stage pulmonary disease, while acute respiratory failure is a common disease among ICU patients. In the early period, following LTx or at the beginning of acute respiratory failure, a protective ventilatory strategy should be applied to reduce ventilator-induced lung injury (VILI). Neurally Adjusted Ventilatory Assist (NAVA) is an assisted ventilation mode in which neural inspiratory activity is monitored through the continuous recording of electrical activity of the diaphragm (EAdi) and then used to coordinate the respiratory support delivered by the ventilator.

NAVA, because of its intrinsic properties (proportionality between respiratory drive and level of assist, prevention of diaphragm atrophy), could allow the aforementioned ventilatory strategy, however it may require the integrity of the pulmonary vagal afferent feedback in order to avoid volutrauma. So, the aim of the study is the evaluation of the physiological relationship between EAdi and tidal volume, driving pressure and mechanical power, at different levels of ventilatory assist, in the absence of pulmonary vagal afferent feedback during early post-operative period after LTx and among critically ill patients affected by acute respiratory failure. Finally, additional parameters will be collected: Pmus, Pocc, transpulmonary pressure etc.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y.o.
* Admission to ICU for post-operative monitoring after LTx or acute respiratory failure needing invasive mechanical ventilation
* Presence of spontaneous breathing activity
* Sedation titrated to a target RASS between 0 and -2
* Written informed consent obtained

Exclusion Criteria:

* Contraindication to nasogastric tube insertion (gastroesophageal surgery in the previous 3 months, gastroesophageal bleeding in the previous 30 days, history of esophageal varices, facial trauma)
* Increased risk of bleeding with nasogastric tube insertion, due to severe coagulation disorders and severe thrombocytopenia ( i.e., INR > 2 and platelets count < 70.000/mm3)
* Severe hemodynamic instability (noradenaline > 0.3 μg/kg/min and/or use of vasopressin)
* Postoperative extracorporeal respiratory support (ECMO)
* Pre-operative reconditioning of the transplanted lungs by means of ex-vivo lung perfusion (EVLP)
* Lung retransplantation
* Failure to obtain a stable EAdi signal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Electrical Activity of the Diaphragm (EAdi) | One hour after the recovery of spontaneous breathing
  Evaluation of the variations of tidal volume Electrical Activity of the Diaphragm in response to different levels of ventilatory assist at different degrees of lung inflation (different Positive End Expiratory Pressure values). Electrical Activity of the Diaphragm (EAdi) (microVolt)
Tidal Volume (mL) and Respiratory rate (Breaths/min) | One hour after the recovery of spontaneous breathing
  Evaluation of the changes in the patient's neural breathing pattern (expressed as mL of Tidal Volume) at different levels of ventilatory assist. Also patient's respiratory rate (Breaths/min) will be evaluated

SECONDARY OUTCOMES:
Driving pressure (DP) | One hour after the recovery of spontaneous breathing, with inspiratory hold manoeuvres
  Evaluation of the variations of DP in response to different levels of ventilatory assist at different degrees of lung inflation. The driving pressure formula is DP = P_plateau - PEEP. It represents the pressure difference between the plateau pressure (P_plateau) and the positive end-expiratory pressure (PEEP) during mechanical ventilation. Unit: mmHg or cmH2O.
Occlusion Pression (Pocc) | One hour after the recovery of spontaneous breathing
  Evaluation of the changes in the patient's respiratory effort (evaluated using Pocc) at different levels of ventilatory assist. The full breath occlusion pressure (Pocc) is the drop in airway-Pressre during a full occluded inspiratory effort. Unit: mmHg or cmH2O.

OTHER OUTCOMES:
PaO2/FiO2 ratio | One hour after the recovery of spontaneous breathing
  Evaluation of the changes in gas exchange, in particular in PaO2/FiO2 ratio, at different levels of ventilatory assist. The emogas analysis was collected from a peripheral artery.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Anaesthesia and Intensive Care, Padua University hospital, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No